CLINICAL TRIAL: NCT03770949
Title: The Feasibility and Acceptability of 3D Printed Orthotics in Children and Adolescents
Brief Title: 3D Printed Orthotics in Children Adolescents
Acronym: PRINT
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Andiamo (Unknown); Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: 233504
Record Dates: First submitted 2018-11-23; First posted 2018-12-10 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2018-11

CONDITIONS: Cerebral Palsy; Ankle Foot Orthosis (AFO)
Keywords: 3-D printing; Children; Adolescents
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 3-D Printed Orthotic (Ankle Foot Orthosis) — Participants will receive a custom individual 3-D printed ankle foot orthosis (AFO).

SUMMARY:
PRINT is a prospective mixed methods study exploring the feasibility and acceptability of providing 3-D printed orthotics specifically an ankle foot orthosis (AFO) to children and adolescents with cerebral palsy.

DETAILED DESCRIPTION:
Children with cerebral palsy often require orthotics or external braces to help them function and to manage or decrease pain, for example an ankle-foot orthoses (AFO). AFOs are orthotics worn on the foot and ankle to maintain the ankle in an optimal position to treat and manage spastic equinus; the AFO can help the child stand, walk, and interact with their peers. AFOs can also prevent muscles and tendons from further tightening and shortening which can contribute to pain, discomfort, loss of range of motion, and disability.

Current thermoplastic orthotic services are expensive, have long wait times and delays in receiving the orthotic which can impact on the fit of the orthotic. An ill-fitting orthosis can lead to impaired skin integrity, pain, further disability, non-compliance with wearing the orthosis, and potential surgery. To overcome these issues technological advances have led to 3-D printed orthotics.

Advantages of 3-D printed orthotics encompass: 0.5-2mm tolerances compared to 10-20mm tolerances in hand manufacturing, lighter materials which decrease the energy needed for mobility such as walking, scanning technology to develop the AFO provides better accuracy, and faster times from scanning to receiving the orthotic. Additionally 3-D printed orthotics allow for more personalisation, and different contextual AFO designs such as a specific AFO for sport.

PRINT is a mixed methods study exploring the experience of children and adolescents with cerebral palsy of receiving and wearing a 3-D printed AFO. Children and adolescents will be recruited from the Royal London Hospital pediatric department. Participants will receive their standard thermoplastic AFO (if the study coincides with their need for a new AFO) and a 3-D printed AFO. Participants will wear their 3-D printed AFO for the duration of the study.

The study aims to explore the participants and their parents/guardians experience of getting the 3-D printed AFO, wearing the AFO, and any impact on their lifestyle or function. This experience will be explored through semi-structured interviews with the child/adolescent and their parent/guardian. The study is also collecting data regarding: fit, comfort, skin integrity, durability of the AFO material, functional outcome measures, and quality of life.

Participants will attend four assessments/visits over the course of the study. Visit 1 encompasses baseline assessments and a painless foot and ankle scan. The foot and ankle scan will be used to develop the 3-D printed AFO. Up to three weeks after visit 1 the participants will attend visit 2 in which they will receive the 3-D printed AFO; the AFO will be assessed for fit and any adjustments will be made. Participants will wear the AFO for three weeks at which point they will attend visit 3. Visit 3 will encompass re-assessment of baseline measures, AFO fit, and assessment skin integrity. If participants have no issues they will continue to wear the 3-D printed AFO for another three weeks. If a participant is having issues or pain resulting from the 3-D printed AFO they will be instructed to wear their standard thermoplastic AFO for the next three weeks if available (remaining in the study). After wearing the AFO for an additional three weeks (three weeks from visit 3), participants will attend the final visit, visit 4. Visit 4 encompasses re-assessment of baseline measures, a resource use questionnaire, and an interview to explore the experience of being fitted for and wearing a 3-D printed AFO.

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents 3-16 years of age with hemiplegia resulting from cerebral palsy who are categorized as either level 1 or level 2 as per the Gross Motor Function Classification for cerebral palsy assessed through a chart review (Children at this level will be able to participate in and complete a walking test)
* Children/adolescents with an identified clinical need for an AFO whose ankle can be held in a corrected position with minimal manual support
* Children/adolescents who are prescribed an AFO for maintenance only assessed through chart review (maintaining joint position)
* Children/adolescents who have previously been prescribed a standard thermoplastic orthotic assessed through chart review

Exclusion Criteria:

* Children/adolescents who require significant amount of manual correction to position their foot
* Children/adolescents with dystonia, spastic diplegia or total body involvement
* Children/adolescents who require bilateral orthotics
* Children/adolescents who require corrective therapy such as serial casting to stretch and reposition the foot and ankle
* Children/adolescents who are participating in another research study that may impact on ankle range of motion or calf muscle length or increase participant burden on parents/participants.
* Children/adolescents weighing more than 62kg as assessed through a chart review
* Children/adolescents that have photo-sensitivity (e.g. epilepsy) assessed through chart review

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents 3-16 years of age who have cerebral palsy, have been previously prescribed and worn a standard thermoplastic AFO for maintenance of ankle position.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Interviews | Interviews will be conducted at visit 4 (9 weeks).
  Semi-structured interviews with participants and their parents/guardians will be completed to explore the experience of being fitted for and receiving a 3-D printed AFO. Interviews will be analyzed using framework analysis, findings will be reported as common themes identified throughout the interviews. Interviews will last approximately 20-30 minutes.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory TM: PedsQL | PedsQL assessed at visit 1 (baseline), 3 (6 weeks), and 4 (9 weeks).
  Self-reported assessment of quality of life will be assessed using the PedsQL. The PedsQL encompasses functional tasks, feelings/emotions, how someone gets on with others, school activities, and participation. The PedsQL has both child report and parent proxy report; there are different questionnaires for different age groups ranging from toddlers to adolescents. Questions are scored on a 5 point Likert scale from 0 to 4; higher scores indicate better health related quality of life.The PedsQL will take approximately 5-10 minutes to complete.
Timed Up and Go Test (TUG) | The TUG will be assessed at visit 1 (baseline), 3 (6 weeks), and 4 (9 weeks).
  The TUG is a functional assessment evaluating sit-stand, ambulation, and turning. The participant starts from a seated position, on 'go' the participant rises from the chair, walks 3 meters turns, walks back to the chair and sits. The test is timed from 'go' to when the participant is back seated in the chair to the nearest centisecond for example 13.46 seconds. This assessment can be done with and with out assistive devices such as walkers or crutches. Faster times are associated with better functional mobility. Three trials will be completed. The TUG will take around 10 minutes to complete.
Range of Motion Assessment | ROM assessment will be completed at visit 1 (baseline), 3 (6 weeks), and 4 (9 weeks).
  Ankle range of motion (ROM) will be assessed using a goniometer, the gold standard in range of motion assessment. The ankle motions assessed are dorsiflexion and plantar flexion to the nearest degree. Three measurement trials will be completed. Ankle range of motion will take approximately 5 minutes to complete.
Resource use/clinical data: previous ankle foot orthoses | The resource use and clinical data will be assessed at visit 4 (9 weeks).
  Participants and their parents/guardians will complete a questionnaire regarding resource use and clinical data such as previous AFO's recording the number of previous AFO's the participant has had.
Resource use/clinical data: Gross Motor Function Classification System | The resource use and clinical data will be assessed at visit 4 (9 weeks) and during screening of patients..
  Participants and their parents/guardians will complete a questionnaire of resource use and clinical data including reporting the participants Gross Motor Function Classification System (GMFCS) which assesses the individuals motor function. The GMFCS level will be the level the individuals scored at their most recent assessment, obtained from participant/guardian report or chart review. GMFCS levels range from I-V; lower levels are associated with higher functioning.
Resource use/clinical data: number of fitting appointments | The resource use and clinical data will be assessed at visit 4 (9 weeks).
  Participants and their parents/guardians will complete a questionnaire of resource use and clinical data including the number of fitting appointments attended to achieve proper AFO fit. This will be done by recording the number of fitting appointments for both the 3-D printed AFO and previous standard AFO's the participant has had.
Resource use/clinical data: compliance wearing the AFO | The resource use and clinical data will be assessed at visit 4 (9 weeks).
  Participants and their parents/guardians will complete a questionnaire regarding resource use and clinical data with questions around compliance with wearing the AFO measured as "yes" compliant with the amount of time prescribed to wear AFO; or "no" not complaint with the amount of team prescribed to wear the AFO and reasons why not complaint (open ended question participant generates their own response).
Resource use/clinical data: skin integrity | The resource use and clinical data will be assessed at visit 4 (9 weeks).
  Participants and their parents/guardians will complete a questionnaire regarding resource use and clinical data with questions around skin integrity (redness, rubbing, skin breakdown) whilst wearing the 3-D printed AFO.
3-D scanning of the lower limb | Visit 1 (baseline assessment)
  The foot and ankle will be scanned using an Artec Eva scanner on a Microsoft Surface 4 tablet with Windows 10. The 3-D scan is what is used to develop and generate the 3-D printed AFO.
  During scanning the tablet camera is used to take a 3-D scan/image of the lower leg, ankle, and foot. The participant does not have to do anything during the 3-D scan. The participant's foot will be placed in the optimal position for the scan and the tablet camera will be moved around the participants' leg and foot to obtain the 3-D image. The 3-D scan is painless and takes around fifteen minutes.
  There are no specific measurements associated with the scanning.

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
n/a no plan to share IPD